CLINICAL TRIAL: NCT06162637
Title: Femoral Neck Locking Plate Vs Multiple Cannulated Cancellous Screws in Treatment of Femoral Neck Fractures in Young Adults: Randomized Controlled Clinical Trial Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eslam Mohamed AHmed (Other)
Responsible Party: Sponsor-Investigator, Eslam Mohamed AHmed, Resident of Orthopaedic department, Sohag University Hospitals, Sohag University
Organization: Sohag University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-11-02MS
Record Dates: First submitted 2023-11-27; First posted 2023-12-08 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Other): grup A with femoral neck fracture will be fixed by femoral neck locking plate
  Interventions: Device: femoral neck locking plate
- B (Other): grup B with femoral neck fracture will be fixed by Multiple cannulated cancellous screws
  Interventions: Device: multiple cannulated cancellous screws

INTERVENTIONS:
Device: femoral neck locking plate — femoral neck fractures fixation by femoral neck locking plate
  Arms: A
Device: multiple cannulated cancellous screws — femoral neck fractures fixation by multiple cannulated cancellous screws
  Arms: B

SUMMARY:
Fracture neck femur are common injuries, especially seen in the elderly in the emergency setting. It is also seen in young patients with high-energy trauma. Immediate diagnosis and management are required to prevent threatening joint complications. Fracture neck femur in young adults is unsolved problem. The preservation of the native hip anatomy and biomechanics is essential in active young adults. Because of the vulnerable blood supply to the femoral part of the hip joint following these fractures, there is a high risk of developing avascular necrosis (AVN) and non-union. Any sort of surgical fixation should aim at preservation the blood supply while securing enough mechanical stability until the fracture unites. Open reduction is indicated in fractures which cannot be anatomically reduced by gentle manipulation. This should be carried out without any delay since this potentially can reduce the incidence of AVN. Treatment of fracture neck femur still controversial. There are several methods for treatment of fracture neck femur as multipe cannulated cancellous screws, locking plate, dynamic hip screw (DHS) with anti-rotational screw, and arthroplasty. There is no internal fixation method superior to another. In this study, we will compare the clinical and radiographic results of femoral neck locking plate vs multiple cannulated cancellous screw in treating femoral neck fractures in young adults.

ELIGIBILITY:
Inclusion Criteria:

* patients (20-55) years
* having unilateral traumatic femoral neck fracture
* idependent walker before trauma without any aids

Exclusion Criteria:

* open fracture
* pathological fracture
* preexisting deformity
* other pelvic or ipsilateral femoral injuries
* renal impairment or were on high dose steroids

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
improvement of pain on the Harris Hip Score (HHS) 6 months post operative | 6 months
  the Harris Hip Score (HHS) is a scale used for evaluating patients following hip fractures. possible scores range for improvement of pain from 44 (no pain) to 0 (totally disabled cripped pain).
Clinical evaluation of gait limping on the Harris Hip Score (HHS) 6 months post operative | 6 months
  the Harris Hip Score (HHS) is a scale used for evaluating patients following hip fractures. possible scores for limping gait range from 11 (none) to 0 (unable to walk).

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Panula J, Pihlajamaki H, Mattila VM, Jaatinen P, Vahlberg T, Aarnio P, Kivela SL. Mortality and cause of death in hip fracture patients aged 65 or older: a population-based study. BMC Musculoskelet Disord. 2011 May 20;12:105. doi: 10.1186/1471-2474-12-105. PMID 21599967
- [Background] Crist BD, Eastman J, Lee MA, Ferguson TA, Finkemeier CG. Femoral Neck Fractures in Young Patients. Instr Course Lect. 2018 Feb 15;67:37-49. PMID 31411399
- [Background] Ly TV, Swiontkowski MF. Treatment of femoral neck fractures in young adults. J Bone Joint Surg Am. 2008 Oct;90(10):2254-66. No abstract available. PMID 18829925
- [Background] Haidukewych GJ, Rothwell WS, Jacofsky DJ, Torchia ME, Berry DJ. Operative treatment of femoral neck fractures in patients between the ages of fifteen and fifty years. J Bone Joint Surg Am. 2004 Aug;86(8):1711-6. doi: 10.2106/00004623-200408000-00015. PMID 15292419
- [Derived] Othman YA, Khalefa AH, Ahmed IM, Ahmed KFE. Femoral neck locking plate versus multiple cannulated screws for femoral neck fractures in young adults: a randomized controlled trial. BMC Musculoskelet Disord. 2025 Aug 18;26(1):799. doi: 10.1186/s12891-025-09019-7. PMID 40826062